CLINICAL TRIAL: NCT02040077
Title: Development and Validation of a Computerized Opioid Overdose Intervention.
Brief Title: Evaluation of a Computerized Opioid Overdose Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Opioid Overdose; R21DA035327 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Computer + Fluency; Computer Only; Treatment as Usual
Keywords: opioid; overdose; OD; opiate; prescription opioids; prescription pain medication; heroin; detoxification; prevention
MeSH Terms: conditions — Drug Overdose | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computer + Fluency (Experimental): Will receive computerized intervention and will be required to periodically demonstrate mastery of information before proceeding to the next module in the computerized intervention.
  Interventions: Behavioral: Computer + Fluency
- Computer Only (Active Comparator): Will receive computerized intervention but will not be required to demonstrate mastery of information as part of the intervention.
  Interventions: Behavioral: Computer Only
- Treatment as Usual (Active Comparator): Will receive publicly available pamphlets that contain same information as the computerized intervention. Will not have access to computerized intervention and will not be required to demonstrate mastery of information as part of the intervention.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Computer + Fluency
  Arms: Computer + Fluency
Behavioral: Computer Only
  Arms: Computer Only
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
Unintentional fatal drug overdose (OD) is now the 2nd leading cause of accidental death in the general population. Fatal OD from opioid analgesics specifically has increased over 400% between 1999 and 2008, and nonfatal overdose occurs at a rate 3-7 greater than fatal OD. Unintentional opioid OD is a public health crisis in several societal populations including drug users, patients being treated for chronic pain, elderly individuals, adolescents, and children. Educational interventions have been developed to increase knowledge regarding opioid OD risk factors, symptoms, and appropriate responses, however no randomized controlled evaluations of these interventions have been conducted. Within-subject evaluations report immediate and sustained increases in participant knowledge and behavior change, yet these programs suffer from limitations that may limit their widespread dissemination. Thus, there is an urgent, critical need to develop an opioid OD educational intervention that can be accessed by a broad audience, and produces immediate and sustained gains in knowledge in an easily administered and cost-effective way. This study will develop a web-based, computerized, interactive, opioid OD education training program that will incorporate multi-media learning components and fluency training to produce knowledge gains. This program will be evaluated using a randomized, controlled comparison of the active intervention against two control interventions. Participants will be recruited from a brief inpatient detoxification (n=75), will receive the intervention immediately upon completing the detoxification (post-treatment), and will complete 2 follow-up visits to evaluate sustained knowledge. The primary outcome will be percent change from baseline on a knowledge test that is administered immediately before and after the intervention, and at a 1 and 3-month follow-up visit. Secondary outcomes will include self-reported behavior change and participant acceptance of the intervention. The study hypothesis is that participants who receive the primary intervention will evidence the largest increase in knowledge gain and retention over time, compared to the control groups. The rationale and public health benefit of this research cannot be understated- this project will make available a brief, empirically-supported intervention that can be administered quickly and easily within hundreds of settings (e.g., treatment centers, prisons and jails, needle exchange centers, primary care offices, schools), and to diverse patient populations (e.g., drug users, chronic pain patients, elderly, student, children, parents). These outcomes are expected to have a positive impact because they will provide cheap, easily-administered intervention strategy that will help reduce the current national epidemic of opioid OD, and will expand the use of computerized interventions to address public health issues more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Age (>18yrs old)
* Past yr diagnosis of opioid dependence
* Recent completion of opioid detoxification

Exclusion Criteria:

* Completion of local overdose prevention programs and/or beta-testing of the computerized intervention
* Physical limitations that will prevent adequate seeing/hearing of the intervention, or from using computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University Bayview Medical Campus, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although the study expected to enroll and randomize 75 participants, an additional participant was randomized into the study - resulting in a final overall sample of 76 randomized participants.
Groups:
- Computer + Questions: Will receive computerized intervention and will be required to periodically answer questions embedded within the program correctly to proceed into the next module.
- Computer Only: Will receive computerized intervention with no embedded questions
- Pamphlet: Receive a printed version of the same intervention
Period: Overall Study
Arm/Group | Computer + Questions | Computer Only | Pamphlet
Started | 27 | 24 | 25
Completed (Completed primary intervention) | 27 | 24 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer + Questions | Computer Only | Pamphlet | Total
Number analyzed (Participants) | 27 | 24 | 25 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.1) | 37.8 (10.6) | 41.9 (14.1) | 39.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 12 | 31
  Male | 15 | 17 | 13 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 24 | 25 | 76

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Gain
Description: The primary outcome is based on performance in the randomized, controlled trial and is change from baseline on a knowledge test that is administered immediately before and after the intervention.
  At the time of the study, no validated scales to assess general information regarding overdose in a true/false manner were available. Therefore the study developed a scale for the purpose of measuring knowledge increase. The scale included 51 items, rated as "true", "false", or "I don't know" (to discourage random guessing from resulting in accurate responses accidentally). The answers to all items were included as part of the intervention content so it was possible for every answer to be learned. The scale was summed together as a single measure of number correct responses (range 0-51) with no subscales. Higher values indicated more correct responses.
Time Frame: Before the intervention (pre-test) and immediately after the intervention (post-test), an average of 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Computer + Mastery: Will receive computerized intervention and will be required to periodically answer questions embedded within the program correctly to proceed into the next module.
Arm/Group | Computer + Mastery | Computer Only | Pamphlet
Number analyzed (Participants) | 27 | 24 | 25
units on a scale
  Pre-Test | 30.6 (5.75) | 30.5 (5.80) | 27.56 (5.94)
  Post-Test | 40.7 (6.22) | 40.5 (6.16) | 36.2 (10.88)

2. Secondary Outcome: Percent Participants Who Would Recommend the Intervention to a Family Member or Friend.
Description: Participant willingness (yes or no) to recommend the intervention to a family member or friend.
Time Frame: Immediately after the intervention (an average of 10 minutes).
Measure: Count of Participants; unit: Participants
Arm/Group | Computer + Mastery | Computer Only | Pamphlet
Number analyzed (Participants) | 27 | 24 | 25
Participants | 27 | 24 | 25

ADVERSE EVENTS:
Groups:
- Pamphlet: Will receive an printed out version of the same intervention.
Arm/Group | Computer + Mastery | Computer Only | Pamphlet
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No